CLINICAL TRIAL: NCT04205253
Title: Is it Possible That Direct Rigid Laryngoscope-related Ischemia-Reperfusion Injury Occurs in the Tongue During Suspension Laryngoscopy as Detected by Ultrasonography: A Prospective Controlled Study
Brief Title: Tongue Depressor-related Ischemia-Reperfusion Injury in Tongue
Status: Completed | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Ozkan Onal, Professor, Selcuk University
Other Study IDs: 2018/330
Record Dates: First submitted 2019-12-17; First posted 2019-12-19 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Side Effect; Ischemia Reperfusion Injury; Edema; Tongue Enlarged
Keywords: tongue; ischemia-reperfusion injury; side effect; edema; suspension laryngoscopy
MeSH Terms: conditions — Reperfusion Injury; Edema; Macroglossia | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study: The first group is the study group. Patients aged 20 years or older and were to undergo suspension laryngoscopy procedure were eligible for inclusion in this group. Tongue areas were measured twice by submental USG. The first measurements (TA1) were done immediately after endotracheal intubation before introducing the rigid direct laryngoscope, whereas the second measurements (TA2) were done after the SL procedure and after removing the rigid direct laryngoscope just before extubation.The difference between TA2 and TA1 (i.e., TA2-TA1) were used to define the occurrence of tongue edema as study group.
  Interventions: Diagnostic Test: Ultrasonography imaging
- Control: The second group was the control group, which included patients who did not need SL and any head and neck procedures.The tongue areas of these patients were measured twice by submental USG as in the study group. The TA1 measurements were done immediately after endotracheal intubation, whereas the TA2 measurements were done at the end of the surgical procedure just before extubation. The difference between TA2 and TA1 (i.e., TA2-TA1) were used to define the occurrence of tongue edema as study group.
  Interventions: Diagnostic Test: Ultrasonography imaging

INTERVENTIONS:
Diagnostic Test: Ultrasonography imaging — This study aimed to evaluate the tongue areas and compare the tongue areas before the implementation of rigid direct laryngoscope and after the rigid direct laryngoscope.

SUMMARY:
This study aimed to detect tongue edema associated with the pressure exerted by a rigid direct laryngoscope by measuring the tongue area using USG in patients undergoing suspension laryngoscopy (SL) procedures.

DETAILED DESCRIPTION:
Suspension laryngoscopy (SL) is a surgical procedure for both diagnostic and therapeutic purposes. In this procedure, a rigid direct laryngoscope is inserted orally, and the tongue and the base of the tongue are compressed.The tongue is an ideal organ for evaluation with ultrasonography. This study aimed to detect the occurrence of tongue edema through ultrasonography examination due to the rigid direct laryngoscope in SL procedures.

ELIGIBILITY:
Study group

Inclusion Criteria:

* Patients aged 20 years or older
* Patients who undergo suspension laryngoscope procedure

Exclusion Criteria:

* refusal to participate
* age of <20 years
* history of syndromal craniofacial abnormalities
* occurrence of tongue masses
* history of craniofacial surgery
* history of burns, trauma or radiotherapy involving the head and neck region
* neurologic disorders and patients with obstructive sleep apnea syndrome (OSAS)
* active inflammation in the head and neck region
* cervical rigidity limiting neck flexion and head extension

Control group

Inclusion Criteria:

Patients aged 20 years or older Patients who did not need suspension laryngoscopy and any head and neck procedures

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 20 years or older who will undergo suspension laryngoscopy procedures or who did not need suspension larygoscopy procedures.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Rate of change in tongue area. | 2018-2019 (6 months)
  This study aimed to measure the change in tongue areas before and after the implementation of rigid direct laryngoscope by using ultrasonography imaging.

SECONDARY OUTCOMES:
Rate of formation in tongue edema. | 2018 (6 months)
  This study aimed to measure the formation of tongue edema due to the rigid direct laryngoscope by using ultrasonography imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Ozkan Onal, Professor, Principal Investigator — Selcuk University
Locations (2):
- Turkey (Türkiye) (2):
  - Selcen Celik, Konya, Selcuklu
  - Selcuk University, Konya, Selcuklu

IPD SHARING:
Plan to Share IPD: No
Individual participant data has been planned to share after publishing as a article in a journal.

REFERENCES:
- [Derived] Onal M, Colpan B, Elsurer C, Bozkurt MK, Onal O, Turan A. Is it possible that direct rigid laryngoscope-related ischemia-reperfusion injury occurs in the tongue during suspension laryngoscopy as detected by ultrasonography: a prospective controlled study. Acta Otolaryngol. 2020 Jul;140(7):583-588. doi: 10.1080/00016489.2020.1743353. Epub 2020 Mar 30. PMID 32223688